CLINICAL TRIAL: NCT03304951
Title: Interventioanl Study of the Sinopsys® Lacrimal Stent in Patients With Moderate to Severe Chronic Rhinosinusitis to Evaluate Safety and Performance for Direct Ethmoid Sinus Saline Irrigation and Ophthalmic Antibiotic/Steroid Delivery
Brief Title: Sinopsys® Lacrimal Stent Indicated for Sinus Irrigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinopsys Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLSEU01
Record Dates: First submitted 2017-02-11; First posted 2017-10-09 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Ethmoid Sinusitis
MeSH Terms: conditions — Ethmoid Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Synopsis® Lacrimal Stent (Experimental): The Sinopsys® Lacrimal Stent is indicated for use in creating a transcaruncular ethmoid sinus access
  Interventions: Device: Sinopsys® Lacrimal Stent

INTERVENTIONS:
Device: Sinopsys® Lacrimal Stent — The Sinopsys® Lacrimal Stent is indicated for use in creating a transcaruncular ethmoid access.
  Other Names: SLS (Sinopsys® Lacrimal Stent)

SUMMARY:
The primary objective is to evaluate clinical data related to the safety and performance of the Sinopsys® Lacrimal Stent.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and performance of the Sinopsys® Lacrimal Stent in the treatment of patients with moderate to severe chronic chronic rhinosinusitis via direct ethmoid sinus saline irrigation and delivery of an ophthalmic antibiotic/steroid drug.

ELIGIBILITY:
Inclusion Criteria:

* Investigator has determined that the potential study subject has moderate to severe chronic rhino sinusitis with ethmoid involvement and has failed medical therapy prior to enrollment.
* Age ≥22 years The potential study subject meets the American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS) criteria for chronic rhino sinusitis (Rosenfeld, et al, 2007)
* 12 weeks or longer of two or more o f the following signs and symptoms:

  * Mucopurulent drainage (anterior, posterior or both)
  * Nasal Obstruction (congestion)
  * Facial pain-pressure-fullness, or
  * Decreased sense of smell and Inflammation si documents by one or more of the following findings:
  * Purulent (not clear) mucus or edema in the middle meatus or ethmoid region
  * Polyps in nasal cavity or the middle meatus, and/or
  * Radiographic imaging showing inflammation of the paranasal sinuses
* SNOT-20 total raw score ≥ 41
* Non-Contrast CT scan (coronal view) confirms depth of olfactory fossa is Keros classification 1or 2 (Gauba, Sleh, Dua, Agarwal, Ell, & Vize, 2006)
* The potential study subject is capable of understanding and executing written informed consent (IC)

Exclusion Criteria:

* Sinus opacification score of ≤ 8 or ≥ 18 measured using the CT derived Lund-Mackay scoring system
* Isolated sinus disease evident on Non-Contrast CT scan that would unlikely to respond to target ethmoid treatment (e.g., isolated sphenoid or frontal disease).
* Polyposis scored as 3 using the Modified Lund-Kennedy Score as follows:

  3 = Polyps completely obstructing the nose
* Prior ocular and/or sinus surgery that alter the boney anatomy or violate/enter the orbit or sinus (i.e. Fess, balloon sinuplasty). Minor procedures such as septoplasty or turbinectomy are not exclusions.
* Prior surgical history, physical exam, nasal endoscopy, and /or imaging studies that suggest significant craniofacial deformity (such as facial anatomic abnormality from surgical intervention, trauma, and congenital or any other cause thus prohibiting adequate placement of the Sinopsys® Lacrimal Stent).
* Presence of a sinonasal encepholocele as determined by Non-Contrast CT scan.
* Presence of active HEENT infection including acute dacryocystitis, with the exception of baseline CRS (Chronic Rhinosinusitis) infection.
* Febrile illness within 2 weeks of procedure and/or active pus from nose.
* Any sign of active ophthalmic disease, infection or inflammation including the presence of severe ocular surface inflammatory disease as determined by ophthalmic and physical exam, which could be exacerbated by the presence of the device.
* Current use of topical medications for the eye to treat an active ophthalmic disease.
* Underlying medical condition that, in the opinion of the Investigator, would place the subject at high risk if PO or IV sedation (MAC or monitored anesthesia care) were used during the procedure.
* Known silicone allergy
* Documented diagnostic history of Cystic Fibrosis
* Documented history of migraines and/or cluster headaches requiring treatment with anti-migraine medication.
* Documented uncontrolled or poorly controlled seasonal or perennial allergies requiring daily anti-allergy oral, nasal or ophthalmic medications.
* Tobacco, marijuana and /or e-vape inhaler use either currently or during the last 6 months
* Documented history of bleeding disorders, for example, von Willebrand's disease or hemophilia.
* Inability to stop thrombolytics or other anti-platelet medication prior to procedure day including but not limited to Coumadin (warfarin) for 5 days, Plavix (clopidogrel) for 3 days, ASA(aspirin)/NSAIDs/fish oil supplements for 10 days, Xeralta® (rivaroxaban) for 24 hours.
* For contact lens wearers, inability to go without contact lenses for at least 10 days postoperatively.
* Known use of any investigational ocular or sinusitis drug(s) or devices within 30 days prior to enrollment.
* Investigator determination that the potential study subject is unable to comply with study procedures and /or follow-up, or provided informed consent.
* Women of childbearing potential who test positive on the study-required urine pregnancy test and who are unwilling to practice a medically acceptable contraception regimen from screening through week 8 visit. Women who are documented as postmenopausal for at least 1 year (> 12 months since last menses) or are surgically sterilized, do not require testing.
* Severe co-morbidity or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, cognitive function, substance abuse, shortened life expectancy, vulnerable patient population, high surgical risk).
* Currently involved in another clinical study where that participation may conflict or interfere with the treatment, follow-up or results of the clinical study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Demonstration of acute procedural/device success | 8 Weeks
  Success defined as successful placement of the Sinopsys® Lacrimal Stent and ability to create and maintain transcaruncular access to the ethmoid sinus with the Sinopsys® Lacrimal Stent for 8 weeks post procedure.
Evaluation of Clinical Success at Week 1, 4 and 8 weeks | 8 Weeks
  Using sterile saline eye drop irrigation and two 10-Day courses of ophthalmic antibiotic/steroid eye drops, defined as improvement in SNOT (Sino-Nasal Outcome Test)-20 compared to baseline.

SECONDARY OUTCOMES:
Compare performance of Screening, 4, and 8 week follow up Modified Lund Kennedy nasal endoscopy scores | 8 Weeks
  Comparison of Endoscopy and CT scores from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Vladan Hrabe, MD, Principal Investigator — Charles University, Pilsen Czech Republic
Locations (1):
- Charles University Faculty of Medicine, Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No